CLINICAL TRIAL: NCT05458739
Title: The ClearCoast™ Magnetic Resonance Outcome Post Marketing Surveillance Study
Brief Title: The ClearCoast™ Magnetic Resonance Outcome PMS Study
Status: Completed | Type: Observational
Sponsor: Clear Cut Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 735CLD Rev.04
Record Dates: First submitted 2022-07-07; First posted 2022-07-14 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment Group: The removed specimen (as part of BCS) is scanned with the ClearCoast MR System.
  Interventions: Device: ClearCoast MR System
- Historical Group: Historical data of patients undergone BCS, under the same eligibility criteria and performed by the same study surgeons, thus minimizing inter-groups and inter-surgeon variability and bias, will serve as a control group for the comparison of the complete resection rate.

INTERVENTIONS:
Device: ClearCoast MR System — The removed specimen is scanned using the ClearCoast MR System.
  Groups: Treatment Group

SUMMARY:
Post Marketing Surveillance (PMS) study. Up to 93 patients undergoing breast conserving surgery will be enrolled in a prospective, single center, non-randomized controlled study, and a corresponding number of historical patients that underwent BCS will serve as the historical control group, accounting for a 1:1 ratio. All study patients and the patients in the historical control group will be required to meet the study eligibility criteria.

BCS will be performed with the routine standard of care (SOC), including intra-operative methods used to improve margin assessment. In addition to SOC process, the main specimen from patients found eligible will be scanned in the ClearCoast™ system. The surgeon will utilize the information from the ClearCoast images in his margin assessments evaluation which includes the diffusion at the surface of a particular aspect (suggesting irregular tissue at the specimen's surface), and decide whether to excise additional tissue. The decision-making process including MR images interpretation and the surgical decisions will be evaluated and documented. Following procedure, routine histopathology examination will be performed accompanied by the ClearCoast optical and parametric maps.

This study is a controlled design, in which subjects previously having undergone BCS by the same surgeons, will serve as the historical control group, comparing the following endpoints:

* Complete surgical re-excision rate
* Total excised breast tissue volume

The study Control group is composed of historical data from patients previously undergone BCS, under the same site SOC surgical practice, practicing surgeons, and study eligible criteria. This allows reducing inter-group variability and bias.

A device operator trained by ClearCut Medical will operate the device throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Women histologically diagnosed with invasive and/or in situ carcinoma of the breast, undergoing primary lumpectomy (partial mastectomy) procedure
2. Age ≥18
3. Patient is willing and capable to provide written Informed Consent Form (ICF)

   Exclusion Criteria:
4. Prior surgical procedure in the same breast within 12 months prior to the surgery date
5. Recurrent breast cancer surgery
6. Neoadjuvant chemotherapy and/or neoadjuvant hormone therapy
7. Previous radiation therapy in the operated breast
8. Pregnancy
9. Lactation
10. Patient has subglandular breast implants in the operated breast
11. moribund patient and/or patient with comorbidities, per principal investigator discretion
12. Participating in any other investigational study for either drug or device which might influence collection of valid data under this study.

    Intraoperative:
13. Specimen undergoing pathological specimen assessment (e.g. by frozen section, imprint cytology or gross assessment by sectioning), resulting in deformation of specimen shape/tissue properties (e.g. Formalin conservation)
14. Specimen dimension is larger than the Tissue container volume (200cc)
15. Inability to define aspect color/orientation and/or margin border

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of women 18 years of age and/or over, who are diagnosed with invasive and/or in situ carcinoma of the breast.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
ClearCoast™ Success rate | 6 months
  the success of the ClearCoast™ system indicating abnormal margins of breast tissue specimen intra-operatively.
  This endpoint compares the proportion of patients that undergo a re-excision surgery following the primary lumpectomy procedure between the two groups.

SECONDARY OUTCOMES:
Secondary Outcome - Re-excision rate | 1 year
  Comparing the percentage of positive margins (%) of the main specimen (as detected by post-operative microscopically as having cancer within 1mm or less of the inked surface) and document which of those positive margins have been addressed by intra-operative re-excision or the absence of further tissue to be re-excised (e.g., undermining the skin or reaching the pectoralis fascia).

CONTACTS AND LOCATIONS:
Locations (2):
- Agaplesion Markus Krankenhaus, Frankfurt, Germany
- Western General Hospital , Breast Unit, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No